CLINICAL TRIAL: NCT02204228
Title: A Post-market Clinical Follow-up Study of the TITAN™ Reverse Shoulder System Used in Primary or Revision Total Shoulder Arthroplasty
Brief Title: TITAN™ Reverse Shoulder System
Status: Terminated | Type: Observational
Why Stopped: Business reasons not related to safety
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-0960-001
Record Dates: First submitted 2014-07-21; First posted 2014-07-30 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis of the Shoulder
Keywords: osteoarthritis; rheumatoid arthritis; post traumatic arthritis; avascular necrosis; severe fractures
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- TITAN™ Reverse Shoulder System (TRS): TITAN™ Reverse Shoulder System (TRS) is a semi-constrained total shoulder construct.
  Interventions: Device: TITAN™ Reverse Shoulder System (TRS)

INTERVENTIONS:
Device: TITAN™ Reverse Shoulder System (TRS) — All patients will be operated on with the TITAN™ Reverse Shoulder System (TRS).

SUMMARY:
The Integra® TITAN™ Reverse Shoulder System (TRS) is a semi-constrained total shoulder construct. When used under the conditions and purposes intended the TRS will relieve pain and restore some functional joint motion to the affected shoulder. The purpose of this study is to assess the short, mid and long term outcomes of the TITAN™ Reverse Shoulder System.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with grossly deficient rotator cuff with severe arthropathy or Subjects with failed joint replacement with grossly deficient rotator cuff
* Subjects with a shoulder joint anatomically and structurally suited to receive the device
* Subjects at least 21 years of age and skeletally mature at the time of surgery
* Subject provided consent to participate in the clinical study (having signed the Informed Consent Form)

Exclusion Criteria:

* Subjects without a functional deltoid muscle
* Subjects with active local or systemic infection
* Subjects with inadequate bone stock in the proximal humerus or glenoid fossa for supporting the components
* Subjects with poor bone quality such as osteoporosis where there could be considerable migration of the prosthesis and/or a chance of fracture of the humerus or glenoid
* Subjects with muscular, neurologic, or vascular deficiencies that compromise the affected extremity
* Subjects with known metal allergies
* Subjects are known to be at risk for lost to follow-up, or failure to return for scheduled visits
* Subjects who are prisoners
* Female subject who are pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require reverse shoulder replacement due to the inclusions below.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Survival (lack of implant component removal or revision) | 2 Year
  Any implant revisions or device related adverse events must be reported as soon as the event is discovered. Assessment of adverse events will occur at each clinic visit.

SECONDARY OUTCOMES:
Efficacy assessed by comparing clinical results after surgery as measured with American Shoulder and Elbow Surgeons Score (ASES) | 2 Year/5 Year/ 7Year/ 10 Year
  Relative change of ASES compared to baseline
Efficacy assessed by comparing clinical results after surgery as measured with EuroQOL-5 Dimension (EQ-5D) score | 2 Year/5 Year/ 7Year/ 10 Year
  Relative change of EQ-5D score compared to baseline
Efficacy assessed by comparing clinical results after surgery as measured with Range of motion (ROM) | 2 Year/5 Year/ 7Year/ 10 Year
  Relative change of ROM compared to baseline
Efficacy assessed by comparing clinical results after surgery as measured with Constant score. | 2 Year/5 Year/ 7Year/ 10 Year
  Relative change of Constant score compared to baseline
Efficacy assessed by comparing clinical results after surgery as measured with Pain Visual Analog Scale (VAS). | 2 Year/5 Year/ 7Year/ 10 Year
  Relative change of Pain Visual Analog Scale (VAS) compared to baseline
Efficacy assessed by comparing clinical results after surgery as measured with SANE (Single Assessment Numeric Evaluation) | 2 Year/5 Year/ 7Year/ 10 Year
  Relative change of SANE compared to baseline
Efficacy assessed by comparing clinical results after surgery as measured with Radiographs | 2 Year/5 Year/ 7Year/ 10 Year
  Outcome after surgery will be evaluated using the Radiographs and comparison with pre-operative data.
Lack of unanticipated device related serious adverse events. | 2 Year/5 Year/ 7Year/ 10 Year
  Any device related adverse events must be reported as soon as the event is discovered. Assessment of adverse events will occur at each clinic visit.
Survival (lack of implant component removal or revision) | 5 Year/7 Year/10 Year
  Any implant revisions or device related adverse events must be reported as soon as the event is discovered. Assessment of adverse events will occur at each clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Karlie Morgan, Study Director — Smith & Nephew, Inc.
Locations (10):
- United States (7):
  - University of Florida, Gainesville, Florida
  - Johns Hopkins University, Columbia, Maryland
  - Mississipi Bone and Joint Clinic, Starkville, Mississippi
  - Active Orthopedics, Glen Ridge, New Jersey
  - Westphal Orthopaedics, Lancaster, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Rothman Institute, Philadelphia, Pennsylvania
- Clinique Bizet, Paris, France
- Hospital de Manacor - Llevant, Manacor, Spain
- Barts Health NHS Trust, London, United Kingdom